CLINICAL TRIAL: NCT02563288
Title: Comparison of Esmolol and Dexmedetomidine on Sympathetic Control During Intracranial Procedures
Brief Title: Esmolol Versus Dexmedetomidine During Intracranial Procedures
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: George Papanicolaou Hospital (Other)
Responsible Party: Principal Investigator, Asouhidou Irene, Consultant anesthesiologist, George Papanicolaou Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GeorgePapanikolaouHospital
Record Dates: First submitted 2015-09-19; First posted 2015-09-30 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Intracranial Aneurysm; Intracranial Neoplasms
Keywords: esmolol; dexmedetomidine; opioids
MeSH Terms: conditions — Intracranial Aneurysm; Brain Neoplasms | interventions — esmolol; Dexmedetomidine; Adrenergic alpha-Agonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esmolol (Active Comparator): Esmolol 500mcg/kg before induction in anesthesia following by 300mcg/Kg/min until extubation.
  Interventions: Drug: Esmolol
- Dexmedetomidine (Active Comparator): Dexmedetomidine 1mcg/Kg following by 0.7mcg/Kg/h until end of surgery.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Esmolol — effect of esmolol on intraoperative sympathetic control and on extubation conditions.
  Other Names: b adrenergic antagonist
  Arms: Esmolol
Drug: Dexmedetomidine — effect of dexmedetomidine on intraoperative sympathetic control and on extubation conditions.
  Other Names: alpha adrenergic agonist
  Arms: Dexmedetomidine

SUMMARY:
Patients undergoing intracranial procedures may experience severe hypertension and tachycardia due to intracranial hypertension and to increased release of adrenaline. Preventing perioperative sympathetic activity is of great importance. A common technique is using b-blockers like esmolol, which effectively block perioperative hemodynamic changes during intracranial surgery. A2 agonists, like Dexmedetomidine-Dex are now being used as a component of a balanced anesthesia during neurosurgical procedures. This study aimed to evaluate whether esmolol or dex attenuates perioperative changes in patients undergoing elective craniotomy with fast track neuroanesthesia.

DETAILED DESCRIPTION:
Patients scheduled for elective craniotomy are randomized to receive Dex 1γ/Kg over 10 minutes following by continuous infusion of Dex 0.7γ/Kg (group D) or esmolol 500mcg/Kg over 5 min following by continuous infusion of 300mcg/Kg/min (group E). Patients in both groups are subjected to a standardized anesthesia comprising of induction with propofol, fentanyl, rocuronium, and maintained with Oxygen-air: 1/1, sevoflurane and bolus fentanyl in order to access the same level of anesthesia (BIS 40-50). The hemodynamic variables at various stages of surgery (HR-heart rate, MAP-Mean arterial pressure) and recovery characteristics are also recorded. It is also performed monitoring of cerebral oximetry (INVOS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA physical status 1-3
* Glasgow Coma Scale:13-15
* Hunt-Hess: 0-3

Exclusion Criteria:

* Patients with ASA physical status >3,
* Body Mass Index (BMI) over 30,
* indication for rapid sequence induction,
* any contraindication for receiving b-blocker,
* Glasgow Coma Scale (GCS) <13,
* history of drug abuse,
* neurologic deficit or preoperatively foreseen delayed extubation,
* preoperative heart rate<45.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Systolic arterial pressure- mean arterial pressure (mmHg) | every 15minutes, starting from the induction in anesthesia through surgery completion and up to first 24 postoperative hours.
  Status of patients during emerge from anaesthesia after intracranial surgery

CONTACTS AND LOCATIONS:
Locations (1):
- George Papanikolaou General Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tanskanen PE, Kytta JV, Randell TT, Aantaa RE. Dexmedetomidine as an anaesthetic adjuvant in patients undergoing intracranial tumour surgery: a double-blind, randomized and placebo-controlled study. Br J Anaesth. 2006 Nov;97(5):658-65. doi: 10.1093/bja/ael220. Epub 2006 Aug 16. PMID 16914460
- [Result] Grillo P, Bruder N, Auquier P, Pellissier D, Gouin F. Esmolol blunts the cerebral blood flow velocity increase during emergence from anesthesia in neurosurgical patients. Anesth Analg. 2003 Apr;96(4):1145-1149. doi: 10.1213/01.ANE.0000055647.54957.77. PMID 12651674